CLINICAL TRIAL: NCT03084666
Title: Remote Ischemic Preconditioning Living Donor Renal Transplant Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Brant Wagener, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F130312023
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: In this study, patients undergoing live donor kidney transplantation will be allocated to the control group or remote ischemic preconditioning group (RIPC). RIPC is the utilization of short periods of ischemia to provide protection of the myocardium or other organ (i.e. kidney) from a subsequent ischemic event.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): The treatment will receive 200 mmHg of pressure from a Zimmer automatic tourniquet system (ATS) for three 5 minute intervals.
  Interventions: Device: Zimmer ATS tourniquet system
- Control Group (Experimental): Our control group will receive 20 mmHg of pressure from a Zimmer automatic tourniquet system (ATS) for three 5 minute intervals.
  Interventions: Device: Zimmer ATS tourniquet system

INTERVENTIONS:
Device: Zimmer ATS tourniquet system — The tourniquet is the same kind that is used in orthopedic surgeries to limit blood loss in arm or leg surgery. It can be inflated to a set pressure for a set amount of time.

SUMMARY:
In this study, patients undergoing live donor kidney transplantation will be allocated to the control group or remote ischemic preconditioning group (RIPC). RIPC is the utilization of short periods of ischemia to provide protection of the myocardium or other organ (i.e. kidney) from a subsequent ischemic event. Before allograft implantation, RIPC will be accomplished in the treatment group donor and control group donor by inducing intermittent extremity ischemia through intermittent inflation of an extremity tourniquet three times for five-minute intervals with five minutes of deflation between inflation periods. The monitored clinical end points will include total urine output following kidney reperfusion over five days, plasma creatinine declination over five days, initiation of dialysis, and development of graft injury. Magnitude of graft injury is the primary endpoint and will be measured using biochemical markers, such as, plasma and urinary concentration of neutrophil gelatinase associated lipocalin (NGAL), interleukin-18 (IL-18), and kidney injury molecule-1 (KIM-1). The sample size calculation is based on a projected difference of NGAL levels between the two study arms. Hall et al reported a mean NGAL level of 49 mg/mL (SD = 37 mg/mL) for a group of patients that had immediate graph function and a mean NGAL level of 248 mg/mL in a group of patients with slow graft function. (which Hall reference is this) Based on these data, a conservative estimate of a mean difference between study groups will be considered 35 mg/mL NGAL. Using these assumptions, an alpha level of 0.05 and 80% power, a sample size of n= 19 per study group will be calculated. By rejecting our null hypothesis, RIPC may serve as a safe, cost-effective protective strategy to prevent allograft injury in the clinical setting of live donor kidney transplantation.

DETAILED DESCRIPTION:
All female patients of childbearing age that qualify for this study will receive a urinary pregnancy test prior to enrollment. Application of a tourniquet will occur after induction of anesthesia and intubation with minimal possibility of causing discomfort as the patient will be anesthetized. The tourniquet will be applied preferably to a leg but an arm will be used if a leg is unavailable. The tourniquet will be inflated for three 5 minute intervals over a 30 minute period of time using the Zimmer A.T.S. 2000 Tourniquet System. Patients will be randomly allocated to one of two groups. The treatment group donor will have the tourniquet inflated on the leg or arm to 200 mmHg. The control group donor will have the tourniquet inflated on the leg or arm to only 20 mmHg. An audible timer will be used to help alert investigators that the tourniquet is in need of deflation after each 5-minute interval. The tourniquet will be removed after the needed 30 minutes of inflation/deflation to prevent inadvertent inflation of the tourniquet. Blood and Urine specimens will be labeled with patient name and medical record number. Urine samples will be taken in the operating room and at 6,12,24,48 hours postoperatively to test for urinary biomarkers at the O'Brien Clinical Research Center. Blood samples for calculation of serum blood urea nitrogen and creatinine will be collected/processed/distributed/stored according to current University of Alabama at Birmingham (UAB) main laboratory guidelines as this test is routinely ordered on renal transplant patients. Urinary biomarker laboratory testing samples will be obtained by a bedside nurse placed in a routine urine sample container and a co-investigator will then bring samples to the laboratory where the samples will be tested for NGAL, KIM-1, and IL-18. Blood samples will be taken daily for the first 5 days. A blood sample will be taken from the patient at 1 month to determine the serum blood urea nitrogen level and the creatinine level. The degree of allograft injury will be assessed by the levels of urinary biomarkers NGAL, IL-18, and KIM-1. Incidence of allograft or transplanted kidney primary malfunction will be based on urine output during the first three days after transplantation, the one month serum creatinine concentration, one month estimated glomerular filtration rate calculated according to diet modification. Additional secondary endpoints include 90-day mortality, length of ICU stay, and length of hospital stay. There is a low probability of tourniquet postoperative pain secondary to time of tourniquet inflation being both intermittent and for a short period of time. Inconvenience includes phone discussions with researchers/coordinators and preoperative discussions addressing risks and benefits of the study. Tourniquets will not be placed on extremities with preexisting arteriovenous fistulas or grafts utilized for hemodialysis. In addition, tourniquets will be placed after oscillometric blood pressure cuff placement for intraoperative anesthesia/surgical monitoring to provide adequate patient blood pressure assessment. The tourniquet will not be placed on the same extremity as the oscillometric blood pressure cuff. The primary investigator or a co-investigator will be present during times of tourniquet inflation. The patient will be assessed for complications immediately after tourniquet removal, in the Post- Anesthesia Care Unit (PACU) , and in the ICU/or step down unit. Finally, patient complication assessment will occur on the transplant floor after effects of anesthesia have completely resolved within 24 hours of tourniquet application. The extremity will also be assessed for injury at the 1-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* > OR = 19 years of age receiving a living donor renal transplant (treatment control group) and their donors (control group donors)

Exclusion Criteria:

* < 19 years of age
* No safe extremity to place tourniquet
* Patients with previous muscle, vascular, or nerve injury to an extremity,
* Patients with only one available extremity that has an arteriovenous fistula
* Patients who are hemodialysis dependent who have not received hemodialysis in the past 4 days
* Paraplegic/quadriplegic patients
* Active pathologic cutaneous lesions on extremities
* Patients with a history of tourniquet pain or complex regional pain syndrome (CRPS)
* Pregnant patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mali Mathru, MD, Principal Investigator — UAB Department of Anesthesiology and Perioperative Medicine
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group Donor: The treatment will receive 200 mmHg of pressure from a Zimmer automatic tourniquet system (ATS) for three 5 minute intervals.
  Zimmer ATS tourniquet system: The tourniquet is the same kind that is used in orthopedic surgeries to limit blood loss in arm or leg surgery. It can be inflated to a set pressure for a set amount of time.
- Control Group Donor: Our control group will receive 20 mmHg of pressure from a Zimmer automatic tourniquet system (ATS) for three 5 minute intervals.
  Zimmer ATS tourniquet system: The tourniquet is the same kind that is used in orthopedic surgeries to limit blood loss in arm or leg surgery. It can be inflated to a set pressure for a set amount of time.
Period: Overall Study
Arm/Group | Treatment Group Donor | Control Group Donor
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group Donor: The treatment will receive 200 mmHg of pressure from a Zimmer ATS tourniquet system for three 5 minute intervals.
  Zimmer ATS tourniquet system: The tourniquet is the same kind that is used in orthopedic surgeries to limit blood loss in arm or leg surgery. It can be inflated to a set pressure for a set amount of time.
- Control Group Donor: Our control group will receive 20 mmHg of pressure from a Zimmer ATS tourniquet system for three 5 minute intervals.
  Zimmer ATS tourniquet system: The tourniquet is the same kind that is used in orthopedic surgeries to limit blood loss in arm or leg surgery. It can be inflated to a set pressure for a set amount of time.
- Total: Total of all reporting groups
Arm/Group | Treatment Group Donor | Control Group Donor | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.3) | 45.7 (11.0) | 45.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 23
  Male | 13 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Biomarkers Measured to Indicate the Magnitude of Graft Injury
Description: Remote ischemic preconditioning (RIPC) will be accomplished in the treatment group donor and control group donor by inducing intermittent extremity ischemia through intermittent inflation of an extremity tourniquet three times for five-minute intervals with five minutes of deflation between inflation periods. The monitored clinical end points will include total urine output following kidney reperfusion. Magnitude of graft injury is the primary endpoint and will be measured using biochemical markers, such as, plasma and urinary concentration of neutrophil gelatinase associated lipocalin (NGAL), interleukin-18 (IL-18), and kidney injury molecule-1 (KIM-1). The sample size calculation is based on a projected difference of NGAL levels between the two study arms.
Time Frame: Baseline
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 20 | 20
pg/ml
  Albumin(in pg/ml) | 17.5 [17.4 to 17.6] | 17.3 [17.2 to 17.8]
  B2M (in pg/ml) | 15.6 [14 to 16.7] | 16.1 [15.4 to 17.3]
  Cystatin C (in pg/ml) | 14.3 [11.6 to 15.5] | 14.9 [14.2 to 15.5]
  EGF (in pg/ml) | 4.7 [4.2 to 5.6] | 5.4 [4.8 to 5.8]
  IGFBP7 (in pg/ml) | 8.8 [8.4 to 9.2] | 9.2 [8.4 to 9.5]
  NGAL (in pg/ml) | 12.2 [11 to 14.4] | 12.9 [12 to 15.4]
  OPN (in pg/ml) | 11.9 [11.2 to 12.1] | 12.6 [11.9 to 13.9]
  TIMP-2 (in pg/ml) | 8.4 [6.3 to 9.4] | 8.1 [7.3 to 10]
  Uromodulin (UMOD) (in pg/ml) | 12.9 [11.8 to 14.3] | 13.6 [12.3 to 14.3]

2. Primary Outcome: Biomarkers Measured to Indicate the Magnitude of Graft Injury
Description: RIPC will be accomplished in the treatment group donor and control group donor by inducing intermittent extremity ischemia through intermittent inflation of an extremity tourniquet three times for five-minute intervals with five minutes of deflation between inflation periods. The monitored clinical end points will include total urine output following kidney reperfusion. Magnitude of graft injury is the primary endpoint and will be measured using biochemical markers, such as, plasma and urinary concentration of neutrophil gelatinase associated lipocalin (NGAL), IL-18, and KIM-1. The sample size calculation is based on a projected difference of NGAL levels between the two study arms.
Time Frame: 6 hours post-operatively
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Biomarkers Measured to Indicate the Magnitude of Graft Injury
Description: as for outcome 2
Time Frame: 12 hours post-operatively
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Biomarkers Measured to Indicate the Magnitude of Graft Injury
Description: as for outcome 2
Time Frame: 24 hours post-operatively
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Biomarkers Measured to Indicate the Magnitude of Graft Injury
Description: as for outcome 2
Time Frame: 48 hours post-operatively
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants That Experienced a Mortality Event
Description: This measure will be a review of those participants that didn't survive this procedure.
Time Frame: From baseline through 90 days
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Length of ICU Stay
Description: The number of days will be counted for their ICU stay
Time Frame: from baseline through 90 days
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Length of Hospital Stay
Description: The entire length of hospital stay will be counted in days
Time Frame: from baseline through 90 days
Population: For both groups this outcome was not measured.
Arm/Group | Treatment Group Donor | Control Group Donor
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events from ischemic preconditioning were monitored for 1 week after treatment/placebo
Arm/Group | Treatment Group Donor | Control Group Donor
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03084666/Prot_SAP_000.pdf